CLINICAL TRIAL: NCT00002923
Title: Phase I Evaluation of KRN5500 (NSC650426)
Brief Title: KRN5500 in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Patricia LoRusso, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065328; U01CA062487 (NIH); P30CA022453 (NIH); WSU-1294; NCI-T96-0004
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — KRN 5500

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KRN5500 (Experimental)
  Interventions: Drug: KRN5500

INTERVENTIONS:
Drug: KRN5500

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to evaluate the effectiveness of KRN5500 in treating patients with metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and toxicities of KRN5500 in patients with solid malignant tumors. II. Characterize the clinical pharmacokinetics of KRN5500 in this patient population. III. Initiate the preliminary evaluation of antitumor activity of KRN5500 in these patients. IV. Determine the recommended Phase II dose of KRN5500.

OUTLINE: This is a dose escalation study. Patients receive KRN5500 IV over 1 hour on days 1-3. Courses repeat every 21 days. Patients with stable disease and partial or complete remission continue treatment for 6 months beyond complete remission. Cohorts of 3 to 6 patients receive escalating doses of KRN5500. The maximum tolerated dose is defined as the dose preceding that at which at least 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study over 9-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven solid malignant tumors with convincing clinical, radiographic or isotopic evidence of dissemination Biopsy proof required in all doubtful cases Must not be eligible for any known regimens or treatments of higher potential efficacy

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: ECOG 0-2 Life Expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT and SGPT no greater than 2 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of acute myocardial infarction within the past 6 months No clinically significant cardiac arrhythmias No New York Heart Association class III or IV disease Other: HIV negative No GI bleeding or bleeding tendency Not pregnant or nursing Effective contraception required for fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Must have recovered from prior biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered At least 6 weeks since prior nitrosourea or mitomycin Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 1997-05; Primary Completion 2000-01 (Actual); Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. LoRusso, DO, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States